CLINICAL TRIAL: NCT06727071
Title: Assessment of Impaired Counterregulatory Hormones and Cardiovascular Risk Using Modern Wearable Sensors in People Living With Type 1 Diabetes.
Brief Title: Using Wearable Sensors To Understand Low Blood Sugar in Type 1 Diabetes
Acronym: Wear WOLF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert L Thomas, Assistant Physician, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 810845
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D; Type 1 Diabetes; Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable Sensor Arm (Other): The intervention is the hyperglycemic clamp. All participants will complete the clamp.
  Interventions: Procedure: Hyperglycemic clamp

INTERVENTIONS:
Procedure: Hyperglycemic clamp — A continuous infusion of 20% dextrose will be maintained throughout the procedure, while a variable rate of insulin infusion will be used to control participants blood glucose level.

SUMMARY:
This is a single-site study using wearable sensor technology (CGM and smartwatch) to better explain low blood sugars in patients living with type 1 diabetes.

Up to 20 participants with T1D will wear a continuous glucose monitor (CGM) and a smartwatch to collect information about hypoglycemia (low blood sugar), heart rate variability (HRV), and sleep for 4 weeks. The main goal is to create a hypoglycemia risk score using wearable sensor metrics that can be easily applied to all patients with T1D to identify those at greater risk of hypoglycemia.

DETAILED DESCRIPTION:
This is a single-site study using wearable sensor technology (continuous glucose monitor [CGM] and smartwatch actigraphy) to stratify hypoglycemia and cardiovascular risk in patients living with type 1 diabetes.

To carry out this research, 20 local participants with Type 1 Diabetes (T1D) will wear CGM and smartwatches to quantify hypoglycemia, heart rate variability (HRV), and sleep actigraphy for 4 weeks. These data will be correlated with counterregulatory hormone levels collected during hyperinsulinemic-hypoglycemic (HHC) clamp. The goal is to create a hypoglycemia risk score using wearable sensor metrics that can be easily applied to all patients with T1D to identify those with impaired counter-regulation in the clinical setting (Aim 1). How hypoglycemia exposure impacts cardiometabolic health in T1D will also be explored.

Participants will complete ambulatory blood pressure monitoring (ABPM), flow mediated dilation (FMD), reactive hyperemia-peripheral artery tonometry (RH-PAT), HRV assessment via wearable smartwatch, and serum inflammatory and coagulation evaluation before and after hyperinsulinemic-hypoglycemic clamp to investigate the effect of hypoglycemia on these cardiovascular (CV) risk factors (Aim 2,3). Subjects will be monitored for 4 weeks prior, and 1 week after hypoglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 75 years old, inclusive, at the time of screening;
2. Females of non-childbearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of childbearing potential must agree to use two methods of contraception during the entire study;
3. Diagnosed with Type 1 diabetes >2-year duration based on clinical history or as defined by the current American Diabetes Association (ADA) criteria;
4. Using hybrid closed loop, standard pump, or multiple daily injections;
5. Able to use a Continuous Glucose Monitoring (CGM) device;
6. A1c > 7% and ≤ 10%:
7. eGFR ≥ 60 mL/min/1.73m²;
8. BMI 18.5-35.0 kg/m2 ;
9. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History or evidence of clinically significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
2. History of pancreatitis, medullary thyroid carcinoma or liver disease:
3. Clinically significant diagnosis of anemia (Hemoglobin < 9 g/dl at screening);
4. Body Mass Index (BMI) < 18.5 kg/m2 and/or weight <50kg;
5. Body Mass Index (BMI) > 35 kg/m2;
6. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed RBCs, platelets or quantities less than 500 mL are allowed at investigator discretion;
7. Current or recent (within 1 month of screening) use of diabetes medications other than insulin; (examples include GLP-1, RA, SGLT-2i, Pramlintide, Metformin);
8. Women who are pregnant or lactating/breastfeeding;
9. Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
10. Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent;
11. Severe hypoglycemic events or DKA within 3 months;
12. Currently using beta-blockers;
13. Adrenal insufficiency diagnosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemic Clamp Epinephrine Response | 160 Minutes
  The change in epinephrine from the start of the clamp to the end as measured in pg/mL.

SECONDARY OUTCOMES:
CGM Time In Range | 4 weeks
  Percent time between 70-180 mg/dL as measured by continuous glucose monitor.
CGM Time Below Range | 4 weeks
  Percent time <70 mg/dL as measured by continuous glucose monitor.
Peripheral Artery Tonometry | 4 weeks
  Change in peripheral artery tonometry as measured by Endo-PAT score.
Brachial Flow Mediated Dilation | 4 weeks
  Change in brachial artery vasodilation as measured by flow mediated dilation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Thomas, MD, PhD, Principal Investigator — UC San Diego
Locations (1):
- University of California, San Diego - ACTRI, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
As the funding for this project is coming from an NIH K12 grant, the data is being used as preliminary data for a K23 submission, so there may not be enough information available to be meaningfully shared.